CLINICAL TRIAL: NCT06932861
Title: Exploratory Study of Personalized mRNA Vaccine in Patients With Refractory Rhabdomyosarcoma
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Xinxin Zhang (Other)
Responsible Party: Sponsor-Investigator, Xinxin Zhang, Director, Department of Otorhinolaryngology - Head and Neck Surgery，Clinical Professor, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRRR Study
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Rhabdomyosarcoma
MeSH Terms: conditions — Rhabdomyosarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vaccine arm (Experimental)
  Interventions: Biological: mRNA Tumor Vaccine Therapy

INTERVENTIONS:
Biological: mRNA Tumor Vaccine Therapy — personalized mRNA vaccines

SUMMARY:
An Exploratory Study on the Use of mRNA Tumor Vaccines in the Treatment of Refractory Rhabdomyosarcoma

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with rhabdomyosarcoma confirmed by pathological or molecular testing;
2. Age ≥ 6 years;
3. No known effective treatment available or no treatment proven to prolong survival with an acceptable quality of life;
4. Expected survival time greater than 6 months;
5. ECOG performance status score of 0-1; -

Exclusion Criteria:

* 1.History of or concurrent with other untreated malignant tumors, except for previously cured basal cell carcinoma of the skin, carcinoma in situ of the cervix, and superficial bladder cancer; 2.History of or current active autoimmune diseases. 3.Has uncontrolled cardiovascular diseases.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Event | From the first administration of the study drug until the occurrence of death, loss to follow-up, withdrawal of informed consent, initiation of a new anti-tumor therapy, or 21 days after the last dose, whichever comes first.

IPD SHARING:
Plan to Share IPD: No